CLINICAL TRIAL: NCT06121895
Title: Evaluation of Differences in Placement Success and Postoperative Complications Between Video Laryngeal Mask Airway and Fastrack Laryngeal Mask
Brief Title: Evaluation of Differences in Video Laryngeal Mask Airway and Fastrack Laryngeal Mask
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf Özgüner, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: AnkaraEtlikYusufOzguner006
Record Dates: First submitted 2023-10-29; First posted 2023-11-08 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: The Device Placement Times; Intubation Times; Postoperative Complications
Keywords: Fastrack Laryngeal Mask; Video Laryngeal Mask
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Video Laryngeal Mask: Patients who are intubated using Video Laryngeal Mask for intubation purposes will be included.
  Interventions: Other: Video Laryngeal Mask
- Fastrack Laryngeal Mask: Patients who are intubated using Fastrack Laryngeal Mask for intubation purposes will be included.
  Interventions: Other: Fastrack Laryngeal Mask

INTERVENTIONS:
Other: Video Laryngeal Mask — Patients who are intubated using Video Laryngeal Mask for intubation purposes will be included.
  Groups: Video Laryngeal Mask
Other: Fastrack Laryngeal Mask — Patients who are intubated using Fastrack Laryngeal Mask for intubation purposes will be included.
  Groups: Fastrack Laryngeal Mask

SUMMARY:
In our study, patients who are intubated using VLM and Fastrack LMA for intubation purposes will be included. The placement times, intubation times, and the number of failed attempts for both devices will be recorded. Additionally, postoperative complications (sore throat, hoarseness, nausea-vomiting, additional antiemetic medication requirements, etc.) will be monitored and recorded.

DETAILED DESCRIPTION:
The 2015 Difficult Airway Society guidelines specify that in cases where an unexpectedly difficult airway is encountered, and the initial intubation attempt is unsuccessful, the insertion of a supraglottic airway device (SAD) is recommended to maintain ventilation and oxygenation, followed by tracheal intubation through the SAD. SAD has been designated as a rescue airway device in difficult airway algorithms and resuscitation guidelines to "buy time." Additionally, SAD is used to maintain airway and anesthesia in surgeries that do not require intubation.

The Video Laryngeal Mask (VLM) is a newly developed type of SAD. With VLM, direct visualization of the glottis is achieved immediately after SAD placement. VLM has a channel that allows for endotracheal tube passage for intubation purposes and provides direct visualization. The Fastrack LMA, on the other hand, possesses all the ventilation features of classic SADs but is designed for blind or fiberoptic-guided tracheal intubations. These devices are used as rescue devices in cases of limited neck extension and difficult airway situations. Both devices are routinely used for ventilation and intubation purposes in patients. The use of these two devices is preferred in patients where neck extension is undesirable or neck movements are restricted for intubation purposes.

In our study, patients who are intubated using VLM and Fastrack LMA for intubation purposes will be included. The placement times, intubation times, and the number of failed attempts for both devices will be recorded. Additionally, postoperative complications (sore throat, hoarseness, nausea-vomiting, additional antiemetic medication requirements, etc.) will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between the ages of 18 and 80.
2. Patients with ASA (American Society of Anesthesiologists) scores I, II, or III.
3. Patients undergoing surgery under general anesthesia in the operating room.

Exclusion Criteria:

1. Patients under 18 years old or over 80 years old.
2. Patients who refuse to participate in the study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Surgical patients undergoing elective surgery and intubated under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Laryngeal Mask Placement times(minute) | 3 minutes after induction of anesthesia
  Laryngeal Mask Placement times(minute)
Intubation times | 3 minutes after induction of anesthesia
  Intubation times
Number of failed attempts | 3 minutes after induction of anesthesia
  Number of failed attempts

SECONDARY OUTCOMES:
Sore throat | 0-2-4-8-12-24 hours postoperatively
  Postoperative complications
Hoarseness | 0-2-4-8-12-24 hours postoperatively
  Postoperative complications
Nausea-vomiting | 0-2-4-8-12-24 hours postoperatively
  Postoperative complications
Need for additional antiemetic medication | 0-2-4-8-12-24 hours postoperatively
  Postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Ozguner, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Varlık Mahallesi, Halil Sezai Erkut Caddesi Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848
- [Result] Van Zundert AAJ, Gatt SP, Van Zundert TCRV, Kumar CM, Pandit JJ. Features of new vision-incorporated third-generation video laryngeal mask airways. J Clin Monit Comput. 2022 Aug;36(4):921-928. doi: 10.1007/s10877-021-00780-3. Epub 2021 Dec 17. PMID 34919170
- [Result] Ferson DZ, Rosenblatt WH, Johansen MJ, Osborn I, Ovassapian A. Use of the intubating LMA-Fastrach in 254 patients with difficult-to-manage airways. Anesthesiology. 2001 Nov;95(5):1175-81. doi: 10.1097/00000542-200111000-00022. PMID 11684987
- [Derived] Ozguner Y, Ozagar UC, Kina SF, Sezgi A, Altinsoy S, Ergil J. Comparison of sacovlm video laryngeal mask-guided intubation and fastrach combined with flexible bronchoscopy-guided intubation -a prospective study. BMC Anesthesiol. 2025 Jul 1;25(1):315. doi: 10.1186/s12871-025-03172-1. PMID 40596865